CLINICAL TRIAL: NCT03829215
Title: Prehospital Cooling of Comatose Patients After Cardiac Arrest With a Non-invasive, Unpowered Core Body Cooling Device (CAERVest Prehospital Cooling)
Brief Title: Prehospital Non-invasive Cooling of Comatose Patients After Cardiac Arrest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: insolvency of the sponsor
Sponsor: Medical University of Vienna (Other)
Collaborators: Bodychillz Ltd (Industry)
Responsible Party: Principal Investigator, Michael Holzer, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.2
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest; Postresuscitation Encephalopathy
Keywords: targeted temperature management; prehospital cooling; cardiac arrest; postresuscitation encephalopathy; resuscitation; heart arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Single centre randomized controlled two arm clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will be comatose on inclusion. Outcome assessor will not be aware of group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAERVest cooling device (Experimental): After checking inclusion and exclusion criteria and immediately after return of spontaneous circulation, the CAERvest device will be filled and placed on the supine patient's chest. A recording esophageal temperature probe will be inserted and connected to the defibrillator. Then the patient will be transported to the Emergency Department.
  After admission to the emergency department, an additional endovascular cooling device will be placed and the patient will be cooled to 33°C for 24 hours with the endovascular cooling device. The CAERvest device will be removed, when a temperature below 34°C is reached.
  Then the patient will be rewarmed at 0.25 °C/h. After rewarming, the temperature will be controlled to be below 37.5°C for until 48 hours after cardiac arrest.
  Interventions: Device: CAERVest cooling device
- Control (No Intervention): After checking inclusion and exclusion criteria and immediately after return of spontaneous circulation, a recording esophageal temperature probe will be inserted and connected to the defibrillator. Then the patient will be transported to the Emergency Department.
  After admission to the emergency department, an endovascular cooling device will be placed and the patient will be cooled to 33°C for 24 hours with the endovascular cooling device.
  Then the patient will be rewarmed at 0.25 °C/h. After rewarming, the temperature will be controlled to be below 37.5°C for until 48 hours after cardiac arrest.

INTERVENTIONS:
Device: CAERVest cooling device — The CAERVest device will be filled and placed on the supine patient's chest immediately after return of spontaneous circulation. After admission to the emergency department, the device will be removed, when a temperature below 34°C is reached.
  Arms: CAERVest cooling device

SUMMARY:
Single centre randomized controlled two arm clinical trial of patients after out of hospital cardiac arrest with return of spontaneous circulation.

The trial objective is to investigate external cooling of cardiac arrest patients after cardiac arrest with the CAERvest cooling device.

After checking inclusion and exclusion criteria and immediately after return of spontaneous circulation, the CAERvest device will be filled and placed on the supine patient's chest. A recording oesophageal temperature probe will be inserted and connected to the defibrillator. Then the patient will be transported to the Emergency Department.

After admission to the emergency department, an additional endovascular cooling device will be placed and the patient will be cooled to 33°C for 24 hours (starting after reaching the target temperature range of under 34°C) with the endovascular cooling device.

Then the patient will be rewarmed at 0.25 °C/h. The CAERvest device will be removed, when a temperature below 34°C is reached.

After rewarming, the temperature will be controlled to be below 37.5°C for until 48 hours after cardiac arrest. After this time point pyrexia (core temperature above 37.5°C) will be treated with common pharmaceutical measures. Sedation, analgesia and relaxation will be discontinued at 36.5°C. Neurologic evaluation will be started not before 72 hours after cardiac arrest with a predefined evaluation protocol. During follow up the following secondary outcomes will be recorded: Survival to hospital discharge, survival to 30 days, survival to 6 months, best neurologic function within 30 days, best neurologic function within 6 months, and quality of life at 6 months.

DETAILED DESCRIPTION:
1 CLINICAL TRIAL PLAN 1.1 Trial Objective The objective of this outcome clinical trial is to evaluate the effectiveness and safety of ultra-early therapeutic hypothermia in cardiac arrest patients using the CAERvest® device.

1.2 Trial Design This clinical trial is a single centre randomized controlled two arm clinical trial. Randomization will be in a 1:1 ratio. The patients will be randomized to a Test Arm (OOH-Cooling; prehospital and in-hospital cooling) or to a Control Arm (Control-Cooling; in-hospital cooling only). The study will include up to 80 patients (40 subjects in each arm).

1.3 Patient Population Subjects will include out of hospital cardiac arrest patients with return of spontaneous circulation, who meet the trial eligibility requirements.

1.4 Clinical Trial Procedures 1.4.1 Patient Screening Patient screening will be conducted by emergency physicians of the emergency medical system (EMS) system of Vienna by help of the Field Supervisor System of the EMS. All out of hospital cardiac arrest, patients with return of spontaneous circulation will be evaluated for inclusion into the trial. The subject's eligibility for the study will be evaluated based on the criteria outlined above in the inclusion/exclusion criteria section.

Enrollment becomes official once eligible subjects meet inclusion/exclusion criteria and the patient is randomized to either Test or Control Arm of the trial.

Subjects may withdraw from the trial at any time at their own discretion with or without reason. Withdrawn subjects will not undergo any additional follow-up, except as desired by mutual agreement of subject and physician. In all cases of withdrawal, the reason(s) for withdrawal (if given) will be recorded upon study termination.

1.4.2 Pre-Cooling Assessment Procedures

Prior to inclusion to the trial, each subject will be assessed for the following:

* Assessment of patient clinical features, signs and symptoms
* Review of Inclusion/Exclusion Criteria
* Patient Randomization
* Availability of an ICU bed at the study centre 1.4.3 Informed Consent The reviewing Medical Ethics Committee (MEC) must review and approve an Informed Consent Form (ICF) specific to this study.

Since this trial is conducted in patients suffering from cardiac arrest, patients will be unconscious and unable to give consent. As it is a prerequisite for cooling and therefore one of the exclusion criteria that the patient has to be comatose on inclusion a formal informed consent will not be possible. According to the law on medicinal devices in Austria, the need for informed consent will be waived. As soon as patients recover and are able to understand the purpose and nature of the trial, they will be informed about their inclusion and informed consent will be sought. If information becomes available that may be relevant to the subject's willingness to continue participating in the trial, the investigator must inform the subject in a timely manner, and a revised written informed consent must be obtained.

The informed consent process (including time and date of discussion), will be documented in the subject's medical record and signed/dated by the individual (investigator or designee) who recorded it. The original signed consent form must be filed in the subject's medical record and a copy of the signed informed consent documentation given to the subject.

In obtaining and documenting informed consent, the investigator must comply with the applicable regulatory requirement(s) and adhere to ICH ( International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use) guideline for good clinical practice (GCP) and the requirements in the Declaration of Helsinki.

1.4.4 Randomization Patients who meet all eligibility criteria for participation will be randomly assigned to either the Test Arm (prehospital + in-hospital cooling) or Control Arm (in-hospital cooling only) in a 1:1 ratio.

Randomization will be done by using a previously prepared sealed envelope. The treating emergency physician at the patient side will open the envelope and act according to the enclosed direction. Subjects will be considered to be enrolled in the Test Arm or Control Arms of the trial when all inclusion and exclusion criteria have been met and randomization assignment has been completed.

1.4.5 Standardized Care Prior to the Cooling Procedure Subjects will receive standard postresuscitation care as part of current clinical practice in the treatment of cardiac arrest (European Resuscitation Council Guidelines 2015). Clinicians will be encouraged to manage the subject in a standardized manner.

For measuring the core temperature an oesophageal temperature probe will be inserted and connected to the defibrillator prehospital immediately after randomization and before start of prehospital cooling (in the Test Arm).

1.4.6 Prehospital Cooling Arm: Temperature Management Protocol and Data Collection Time Points Treatment with therapeutic hypothermia will begin immediately after randomization and placement of the oesophageal temperature probe with the CAERvest® device. The device will be filled with the provided fluid and then be placed on the patient's chest. After admission to the emergency department cooling will then be continued as soon as possible with an endovascular cooling device (Thermogard XP®, Zoll, San Jose, USA) set at a temperature of 33.0 °C. The subject's core temperature will then be further measured by an oesophageal temperature probe connected to ICU-Monitor and the Thermogard XP®. The cooling device will be removed, when a temperature below 34°C is reached. Cooling will be maintained for 24 hours (starting after reaching the target temperature range of under 34°C) and will be followed with active rewarming (at 0.25 °C/h) to attain normothermia (36.0 °C). After rewarming, the temperature will be controlled to be below 37.5°C for 48 hours after cardiac arrest. After this time point pyrexia will be treated with common pharmaceutical measures. Sedation, analgesia and relaxation will be discontinued earliest at a core temperature of 36.5°C.

1.4.7 Control Arm: Temperature Management Protocol and Data Collection Time Points Treatment with therapeutic hypothermia will begin as soon as possible after admission to the emergency department with an endovascular cooling device (Thermogard XP®) set at a temperature of 33.0 °C. The subject's core temperature will be measured via an oesophageal temperature probe connected to ICU-Monitor and the Thermogard XP®. Cooling will be maintained for 24 hours (starting after reaching the target temperature range of under 34°C) and will be followed with active rewarming (at 0.25 °C/h) to attain normothermia (36.0 °C). After rewarming, the temperature will be controlled to be below 37.5°C for 48 hours after cardiac arrest. After this time point pyrexia will be treated with common pharmaceutical measures. Sedation, analgesia and relaxation will be discontinued earliest at a core temperature of 36.5°C.

1.4.8 Follow-up Subjects enrolled in the study will undergo defined follow up time points after return of spontaneous circulation (ROSC). At 6h, 12h, 24h, 44-52h, 68-76h, 6-8days, 1 month and 6 months data will be collected according to the Utstein-style guidelines (data on details of the cardiac arrest, baseline demographic data, Pittsburgh Brain Stem Score, Cerebral Performance Category score, and Overall Performance Category score). At specific time points, blood samples for laboratory examinations and blood gases will be obtained as a standard procedure after cardiac arrest. At 6 months, quality of life will be assessed with the Short Form (36) Health Survey (SF-36) and the Health Utilities Index Mark 3 system (HUI3) by researchers blinded to study allocation.

1.4.9 Patient Withdrawal and Discontinuation The term "patient withdrawal" refers to the patient deciding to terminate their participation in the trial. The term "discontinuation" refers to the physician deciding that the patient will not continue trial participation as defined below.

A subject has the right to withdraw from the trial at any time and for any reason without prejudice to his or her future medical care by the physician or the institution. Trial withdrawal by a subject specifically means withdrawal of consent from further participation in the trial. Subjects who withdraw consent after enrollment will be evaluated to the time of withdrawal, and withdrawal of consent precludes any further trial related treatment or data collection. If possible, a complete, final physical examination should be performed on all subjects who withdraw from the trial. At a minimum, every effort should be made to document subject outcome at the time of trial withdrawal.

A subject may be discontinued from the clinical investigation for the following reasons:

* Any unanticipated adverse reaction which is, in the opinion of the Investigator, related to the treatment and will endanger the well-being of the patient if treatment is continued;
* Development of any illness(es), infection or condition(s) that might interfere with the Clinical Investigational Plan;
* Non-compliance with the clinical investigation procedures deemed by the Investigator to be sufficient to cause discontinuation;
* Any problem deemed by the Investigator to be sufficient to cause discontinuation.

Investigator will treat all subjects discontinued from the investigation due to an unanticipated adverse reaction, directly related to the investigation, until the reaction resolves.

Investigator will not replace subjects who have withdrawn from the clinical investigation if they have received the investigational device. If possible, Investigator will perform any procedures or assessments planned for the subject at the time of withdrawal.

All subjects are expected to continue in the trial through the final follow-up assessment or until BodyChillz Ltd notifies the Investigator in writing, that further follow-up is no longer required, except in the event of death or upon the subject's request for early withdrawal from the clinical trial.

1.4.10 Patient Lost to Follow-up The investigator will attempt to contact a subject at least three times prior to designating them as lost-to-follow-up subjects. The investigator will document the date and type of attempted communication. The investigator will complete and sign the Study Exit Form when a subject is lost to follow-up.

1.4.11 Early Termination of the Clinical Investigation Both the Sponsor and Investigator reserve the right to terminate the clinical investigation at any time. If necessary, and after review and consultation with Principal Investigator, Sponsor will make a final determination on whether to terminate the study.

A clinical investigation or Investigator may be terminated for any of the following reasons, or for reasons not listed that affect patient safety or integrity of the trial:

* Unsatisfactory rate of patient enrollment or compliance to eligibility criteria.
* Repeated noncompliance with the investigational plan.
* Inaccurate, incomplete, and/or untimely submission of data.
* Inadequate accountability of the investigational device. The sponsor may terminate this trial if there are new, previously unknown adverse events related to the device or cooling procedure, deaths, serious adverse events / adverse events exceeding those reported as related to device/cooling procedures in previous trials. The sponsor will make the final determination on whether to terminate the study.

1.4.12 Trial Exit The Trial Exit Form (CRF) should be completed at the time a subject is exited from the trial. A subject will be considered to have exited from the trial for any of the following reasons.

* Subject completes follow-ups required by the investigational plan.
* Subject dies.
* Subject requests to be withdrawn.
* Physician requests that patient be withdrawn to protect the welfare of the patient.
* Patient is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Witnessed cardiac arrest
3. Restoration of spontaneous circulation
4. All Primary rhythms
5. Cardiac arrest of presumed cardiac origin

Exclusion Criteria:

1. Hypothermia (< 34 °C) on screening
2. Comatose prior to cardiac arrest due to central nervous system depressant drugs
3. CPC higher than 2 prior to cardiac arrest
4. Known pregnancy
5. Glasgow coma scale (GCS) > 8 at screening
6. Known malignancy e.g. terminal illness (pre-cardiac arrest life expectancy of < 6 months due to underlying medical conditions or pre-existing co-morbidities.)
7. Follow up unlikely to be possible
8. Patients already randomized to a clinical trial
9. The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia, sickle cell anaemia, or will refuse blood transfusions
10. The patient is a vulnerable subject, for instance, a person in detention (i.e., prisoner or ward of the state)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cooling rate | 4 hours
  Significant reduction of oesophageal temperature with the CAERvest cooling device compared to the control group at start of the endovascular cooling device, calculated as the difference in core temperature at start of second cooling device and initial core temperature by time.

SECONDARY OUTCOMES:
Earlier achievement of target temperature | 4 hours
  Achievement of target temperature is defined as the time point when the patient reaches a temperature below 34°C. The time interval between ROSC and this time point will be reported.
Ease of use and operator experience with the cooling device | 4 hours
  This will be assessed by the means of an operator survey performed immediately on admission of the patient. The following items will be recorded:
  Problems with unpacking device, fluid Leakage post activation, problems with connecting reservoir, problems with Air Lock, problems with CAERVest placement, interfering of cardiopulmonary resuscitation due to device, dry chemical leakage, problems with defibrillation.
Survival to hospital discharge | 14 days
Survival to 30 days | 30 days
Survival to 6 months | 6 months
Best neurologic function within 30 days | 30 days
  Measured by CPC (Cerebral Performance Category) score. CPC scores are defined as follows: CPC-1 is conscious and normal, without disability, CPC-2 is conscious with moderate disability, CPC-3 is conscious with severe disability, CPC-4 is a comatose or vegetative state and CPC-5 is defined as death.
Best neurologic function within 6 months | 6 months
  Measured by CPC (Cerebral Performance Category) score. CPC scores are defined as follows: CPC-1 is conscious and normal, without disability, CPC-2 is conscious with moderate disability, CPC-3 is conscious with severe disability, CPC-4 is a comatose or vegetative state and CPC-5 is defined as death. The best achieved score within 6 months will be recorded.
Quality of life at 6 months | 6 months
  Measured by HUI-3 (Health Utilities Index Mark 3). In HUI-3, utility values range from -0.36 to 1.00. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. To account for the fact that some health states are identified by the general public as being worse than death, the score could also be negative. To calculate a health utility score, health states for each response are converted using a look-up table and mathematical formula. Each attribute and level has a corresponding coefficient value to be input into the formula to calculate health utility.
Quality of life at 6 months | 6 months
  Measured by the SF-36 (Short Form (36) Health Survey). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 14 days
  The occurrence of the following adverse events within 14 days after inclusion will be recorded: Skin damage / cold burns, death, acute renal failure, clinically relevant shivering (BSAS ≥ 2) that cannot be controlled by the antishivering medication regimen, dysrhythmia [ventricular tachycardia, ventricular fibrillation or atrial fibrillation requiring intervention, bradycardia (HR ≤ 40 bpm, block)], hyperglycemia / hypoglycaemia, hyperkalaemia / hypokalemia, infection, multi-system organ failure, overcooling (temperature <31.0°C for ≥ 20 continuous minutes), pancreatitis, thrombocytopenia and seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holzer, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamarainen A, Virkkunen I, Tenhunen J, Yli-Hankala A, Silfvast T. Prehospital therapeutic hypothermia for comatose survivors of cardiac arrest: a randomized controlled trial. Acta Anaesthesiol Scand. 2009 Aug;53(7):900-7. doi: 10.1111/j.1399-6576.2009.02015.x. Epub 2009 Jun 3. PMID 19496762
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Holzer M, Bernard SA, Hachimi-Idrissi S, Roine RO, Sterz F, Mullner M; Collaborative Group on Induced Hypothermia for Neuroprotection After Cardiac Arrest. Hypothermia for neuroprotection after cardiac arrest: systematic review and individual patient data meta-analysis. Crit Care Med. 2005 Feb;33(2):414-8. doi: 10.1097/01.ccm.0000153410.87750.53. PMID 15699847
- [Background] Uray T, Mayr FB, Stratil P, Aschauer S, Testori C, Sterz F, Haugk M. Prehospital surface cooling is safe and can reduce time to target temperature after cardiac arrest. Resuscitation. 2015 Feb;87:51-6. doi: 10.1016/j.resuscitation.2014.10.026. Epub 2014 Nov 28. PMID 25447355
- [Background] Nielsen N, Wetterslev J, Cronberg T, Erlinge D, Gasche Y, Hassager C, Horn J, Hovdenes J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher M, Wise MP, Aneman A, Al-Subaie N, Boesgaard S, Bro-Jeppesen J, Brunetti I, Bugge JF, Hingston CD, Juffermans NP, Koopmans M, Kober L, Langorgen J, Lilja G, Moller JE, Rundgren M, Rylander C, Smid O, Werer C, Winkel P, Friberg H; TTM Trial Investigators. Targeted temperature management at 33 degrees C versus 36 degrees C after cardiac arrest. N Engl J Med. 2013 Dec 5;369(23):2197-206. doi: 10.1056/NEJMoa1310519. Epub 2013 Nov 17. PMID 24237006
- [Background] Arrich J, Holzer M, Havel C, Mullner M, Herkner H. Hypothermia for neuroprotection in adults after cardiopulmonary resuscitation. Cochrane Database Syst Rev. 2016 Feb 15;2(2):CD004128. doi: 10.1002/14651858.CD004128.pub4. PMID 26878327
- [Background] Uray T, Malzer R; Vienna Hypothermia After Cardiac Arrest (HACA) Study Group. Out-of-hospital surface cooling to induce mild hypothermia in human cardiac arrest: a feasibility trial. Resuscitation. 2008 Jun;77(3):331-8. doi: 10.1016/j.resuscitation.2008.01.005. Epub 2008 Mar 7. PMID 18314248
- [Background] Kim F, Olsufka M, Longstreth WT Jr, Maynard C, Carlbom D, Deem S, Kudenchuk P, Copass MK, Cobb LA. Pilot randomized clinical trial of prehospital induction of mild hypothermia in out-of-hospital cardiac arrest patients with a rapid infusion of 4 degrees C normal saline. Circulation. 2007 Jun 19;115(24):3064-70. doi: 10.1161/CIRCULATIONAHA.106.655480. Epub 2007 Jun 4. PMID 17548731
- [Background] Bernard SA, Smith K, Cameron P, Masci K, Taylor DM, Cooper DJ, Kelly AM, Silvester W; Rapid Infusion of Cold Hartmanns Investigators. Induction of prehospital therapeutic hypothermia after resuscitation from nonventricular fibrillation cardiac arrest*. Crit Care Med. 2012 Mar;40(3):747-53. doi: 10.1097/CCM.0b013e3182377038. PMID 22020244
- [Background] Kim F, Nichol G, Maynard C, Hallstrom A, Kudenchuk PJ, Rea T, Copass MK, Carlbom D, Deem S, Longstreth WT Jr, Olsufka M, Cobb LA. Effect of prehospital induction of mild hypothermia on survival and neurological status among adults with cardiac arrest: a randomized clinical trial. JAMA. 2014 Jan 1;311(1):45-52. doi: 10.1001/jama.2013.282173. PMID 24240712
- [Background] Bernard SA, Smith K, Cameron P, Masci K, Taylor DM, Cooper DJ, Kelly AM, Silvester W; Rapid Infusion of Cold Hartmanns (RICH) Investigators. Induction of therapeutic hypothermia by paramedics after resuscitation from out-of-hospital ventricular fibrillation cardiac arrest: a randomized controlled trial. Circulation. 2010 Aug 17;122(7):737-42. doi: 10.1161/CIRCULATIONAHA.109.906859. Epub 2010 Aug 2. PMID 20679551
- [Background] Kamarainen A, Virkkunen I, Tenhunen J, Yli-Hankala A, Silfvast T. Induction of therapeutic hypothermia during prehospital CPR using ice-cold intravenous fluid. Resuscitation. 2008 Nov;79(2):205-11. doi: 10.1016/j.resuscitation.2008.07.003. Epub 2008 Sep 21. PMID 18809236
- [Background] Arrich J, Holzer M, Havel C, Warenits AM, Herkner H. Pre-hospital versus in-hospital initiation of cooling for survival and neuroprotection after out-of-hospital cardiac arrest. Cochrane Database Syst Rev. 2016 Mar 15;3(3):CD010570. doi: 10.1002/14651858.CD010570.pub2. PMID 26978162